CLINICAL TRIAL: NCT00889239
Title: Clinical Performance and Wear Mechanism of Hot-Pressed Ceramic Crowns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Thailand Research Fund (Other)
Responsible Party: Principal Investigator, Kallaya Suputtamongkol, Dr., Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRG 4780066
Record Dates: First submitted 2009-04-25; First posted 2009-04-28 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: Ceramic and Dental Enamel Wear
Keywords: ceramic; wear rate; opposing enamel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): ceramic crown
  Interventions: Other: lithia-disilicate-based crown

INTERVENTIONS:
Other: lithia-disilicate-based crown — all-ceramic crown
  Other Names: ceramic crown

SUMMARY:
The objectives of this study are to characterize the clinical performance and wear mechanisms of all-ceramic posterior crowns. The wear rate of all-ceramic crowns and opposing enamel in selected patients will be quantified. The relationship of each subject's maximum clenching force and wear rate will also be analyzed.

DETAILED DESCRIPTION:
High strength ceramics have been used in dentistry for constructing fixed partial denture. Their advantages are their acceptable fracture resistance, excellent biocompatibility, moderate opacity, etc. Because the increase in demand for more esthetic restoration, various ceramic materials have been used as a core material for several all-ceramic systems. Their properties have been investigated extensively in many in vitro studies. Currently, there are not much results regarding clinical performance and wear mechanism of ceramic-based prosthesis and more information are required for future research.

ELIGIBILITY:
Inclusion Criteria:

* Occlusion: At least 20 remaining teeth for each patient, and at least one posterior endodontically treated tooth with natural opposing teeth
* Bruxism: No evidence based on an intraoral examination
* Dental history: No evidence of either moderate or severe periodontal disease
* Medical history: Good to excellent general health

Exclusion Criteria:

* Periodontal status: Pocket depth greater than 4 mm
* Occlusion:

  * Evidence of bruxism or excessive biting or clenching force
  * Abutment tooth that opposes a removable partial denture
  * Abutment tooth for fixed partial dentures
  * Gingival recession of an abutment tooth more than 1 mm from the cementoenamel junction
  * Tooth with first or second degree of tooth mobility
  * Tooth with extensive carious lesions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2004-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Clinical performance | 5 years

SECONDARY OUTCOMES:
wear rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kallaya Suputtamongkol, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Dentistry, Mahidol University, Bangkok, Thailand